CLINICAL TRIAL: NCT01590849
Title: Assessment of Autonomic Tone in Normotensive Women Using Combined Hormonal Oral Contraceptive Containing Drospirenone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Marcelo Gil Nisenbaum, post graduate and contributor to the medical clinic for family planning of the Department of Gynecology of Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: nisenbaum1
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Contraceptive Affecting the Autonomic Nervous System; Contraceptive Affecting Blood Pressure
Keywords: contraceptive agents; autonomic nervous system; blood pressure; risk
MeSH Terms: interventions — Contraceptive Agents; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No hormonal contraception (No Intervention)
- Hormonal Contraceptive (Active Comparator): healthy women, users of COC containing 20 mcg EE and 3 mg DRSP (Yaz®), 24 days of active pills, 4 days of pill-free interval (n=40).
  Interventions: Drug: Contraceptives, Oral, Combined (Yaz®)

INTERVENTIONS:
Drug: Contraceptives, Oral, Combined (Yaz®) — After a counseling session concerning the advantages, disadvantages and side effects of contraceptive methods (COC or nonhormonal methods), the volunteers were divided into two study groups according to the method they chose to use as follows:
  * Case group: healthy women, users of COC containing 20 mcg ethynil estradiol and 3 mg drospirenone , 24 days of active pills, 4 days of pill-free interval (n=40).
  * Control group: healthy women, users of nonhormonal methods of contraception (condoms or copper IUD) (n=40).
  Subjects were tested once before the introduction of the contraceptive method and again after 6 months of its use.
  Other Names: Brand Name in Brazil - (Yaz®)
  Arms: Hormonal Contraceptive

SUMMARY:
The use of combined oral contraceptives has been associated with increased risk of adverse cardiovascular events. The exact mechanism by which these drugs exert this influence is uncertain. It is possible that changes in autonomic nervous system are involved. The objective of these study was to evaluate the effect of the use of a contraceptive containing 20 mcg of ethinyl estradiol and 3mg of drospirenone in the autonomic nervous system in healthy women. Few studies have been conducted in the field of hormonal contraception and evaluation of the autonomic nervous system work and no prospective, controlled study was published so far. These study will be the first.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years old
* no use of hormonal contraceptives for at least 6 months before the study
* need for contraceptive method
* willingness to participate in the study

Exclusion Criteria:

* positive pregnancy test
* category 3 or 4 classification on WHO's Medical Eligibility Criteria for Contraceptive
* smoking
* obesity
* fasting glucose above 100 mg/dL
* abnormalities in lipid profile
* use of other medications

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
combined hormonal oral contraceptive with drospirenone and its influence on the autonomic nervous system | six months after the intervention
  The participants in this study will be 80 healthy women. After a counseling session concerning the advantages, disadvantages and side effects of contraceptive methods (COC or nonhormonal methods), the volunteers were divided into two study groups according to the method they chose to use as follows:
  * Case group: healthy women, users of COC containing 20 mcg EE and 3 mg DRSP (Yaz®)(n=40).
  * Control group: healthy women, users of nonhormonal methods of contraception (condoms or copper IUD) (n=40).
  The acquisition of autonomic parameters will be performed through the device Finometer.

SECONDARY OUTCOMES:
combined hormonal oral contraceptive with drospirenone and its influence on blood pressure | six month after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo G Nisenbaum, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Marcelo Gil Nisenbaum, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Carter JR, Klein JC, Schwartz CE. Effects of oral contraceptives on sympathetic nerve activity during orthostatic stress in young, healthy women. Am J Physiol Regul Integr Comp Physiol. 2010 Jan;298(1):R9-R14. doi: 10.1152/ajpregu.00554.2009. Epub 2009 Oct 14. PMID 19828840
- [Background] Minson CT, Halliwill JR, Young TM, Joyner MJ. Sympathetic activity and baroreflex sensitivity in young women taking oral contraceptives. Circulation. 2000 Sep 26;102(13):1473-6. doi: 10.1161/01.cir.102.13.1473. PMID 11004135